CLINICAL TRIAL: NCT06483386
Title: Pyrotinib and Subcutaneous Preparation of Trastuzumab Combined With Capecitabine Neoadjuvant Therapy for HER2+Single Arm Phase II Multicenter Study of Breast Cancer
Brief Title: Pyrotinib and Subcutaneous Preparation of Trastuzumab Combined With Capecitabine Neoadjuvant Therapy for HER2+ Study of Breast Cancer
Status: Not yet recruiting | Phase: Phase 2 | Type: Interventional
Sponsor: Tianjin Medical University Cancer Institute and Hospital (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: Tianjin Cancer Hospital .
Record Dates: First submitted 2024-06-12; First posted 2024-07-03 (Actual); Last update posted 2024-07-03 (Actual); Status verified 2024-06

CONDITIONS: Breast Cancer
MeSH Terms: conditions — Breast Neoplasms | interventions — pyrotinib; Capecitabine

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Treatment group (Experimental): Pyrotinib Maleate Tablets: Continuously administered from day 1 of the first course of treatment, 400 Mg/day, orally administered within 30 minutes after breakfast Trastuzumab: Subcutaneous injection, 600mg, d1, q3w Capecitabine: oral, 1000 mg/m2
  , bid d1-14,q3w Premenopausal goserelin 3.6mg once every 28 days
  Interventions: Drug: Pyrotinib and Subcutaneous preparation of trastuzumab combined with capecitabine

INTERVENTIONS:
Drug: Pyrotinib and Subcutaneous preparation of trastuzumab combined with capecitabine — Pyrotinib and Subcutaneous preparation of trastuzumab combined with capecitabine

SUMMARY:
Objective: To explore the efficacy and safety of Pyrotinib, trastuzumab subcutaneous preparation and capecitabine neoadjuvant therapy for early HER2+breast cancer.

Administration method: 6 cycles throughout the entire process:

Pyrotinib Maleate Tablets: Continuously administered from the first day of the first course of treatment, 400 Mg/day, orally administered within 30 minutes after breakfast Trastuzumab: Subcutaneous injection, 600mg, d1, q3w Capecitabine: oral, 1000 mg/m2, bid d1-14, q3w Premenopausal goserelin 3.6mg once every 28 days

DETAILED DESCRIPTION:
Inclusion Criteria :1. Age: Female first-time patients aged 18 and above; 2. Pathological examination confirmed HER2 positive invasive breast cancer; (HER2 positive definition) Further application of in situ hybridization (ISH) for immunohistochemistry (IHC) 3+or IHC 2+ HER2 gene amplification, regardless of hormone receptor status (ER and PR); According to the eighth edition of AJCC, the staging is T1c-2N0-1M0, and according to Recipe 1.1, there are At least one measurable lesion; 4. ECOG PS: 0-1 points; 5. The main organ function is normal, which meets the following standards:

1. The standard for blood routine examination must comply with (no blood transfusion or blood products within 14 days, no use of G-CSF)

   Correction of other hematopoietic stimulating factors:

   Hb≥100g/L； ANC ≥ 1.5 × 10 9/L; PLT ≥ 100 × 10 9/L;
2. Biochemical examination must meet the following standards:

   TBIL ≤ 1 × ULN; ALT, AST ≤ 1.5 × ULN; ALP ≤ 2.5 × ULN; BUN and Cr ≤ 1.5 × ULN;
3. Cardiac ultrasound:

Left ventricular ejection fraction (LVEF) ≥ 55%; 6. Women of childbearing age must undergo a pregnancy test (serum) within 7 days before enrollment, and the result is negative Sexual and willing to use appropriate medication during the trial period and within 8 weeks after the last administration of the investigational drug The method of contraception; 7. The subjects voluntarily joined this study, signed an informed consent form, had good compliance, and cooperated with follow-up.

Exclusion criteria:

Those who are unable to participate in the clinical study under any of the following circumstances:

1. Have received any form of anti-tumor treatment in the past (chemotherapy, radiotherapy, molecular targeted therapy,...) Endocrine therapy, etc;
2. Simultaneously receiving any other anti-tumor treatment;
3. Bilateral breast cancer, inflammatory breast cancer or occult breast cancer;
4. breast cancer not confirmed by histopathology;
5. Other malignant tumors have appeared within the past 5 years, except for cured cervical cancer in situ;
6. Severe dysfunction of important organs such as heart, liver, and kidney;
7. Unable to swallow, chronic diarrhea, and intestinal obstruction, there are various factors that affect medication administration and absorption Factors;
8. Participated in clinical trials of other drugs within 4 weeks prior to enrollment;
9. Individuals with a known history of allergies to the drug components of this protocol; History of immunodeficiency, including HIV Test positive, HCV, active hepatitis B, or other acquired diseases Natural immunodeficiency disease or a history of organ transplantation;
10. Have ever suffered from any heart disease, including: (1) those that require medication or have clinical significance Arrhythmias; (2) Myocardial infarction; (3) Heart failure; (4) Any researcher Other heart diseases deemed unsuitable for participation in this trial;
11. Pregnant and lactating female patients with fertility and positive baseline pregnancy test results Female patients of childbearing age who are unwilling to take effective contraceptive measures throughout the entire trial period Female patients;
12. According to the researcher's judgment, there is a serious threat to patient safety or an impact on patient completion of the study The accompanying diseases studied (including but not limited to severe hypertension that cannot be controlled by medication, severe Diabetes, active infection, etc.);
13. Have a clear history of neurological or psychiatric disorders, including epilepsy or dementia. Researchers believe that Any other circumstances in which the patient is not suitable to participate in this study.

Termination of study standard:

1. Completed treatment according to regulations;
2. Imaging evidence indicates progression of the disease;
3. After dose adjustment, the subjects still cannot tolerate toxicity; During the research process, pregnancy events occurred in the subjects;

5. The subject withdraws their informed consent and requests withdrawal; 6. Other situations where the researcher deems it necessary to withdraw from the study.

efficacy indicators:

Main efficacy indicators:

tpCR

Secondary efficacy indicators:

1. pCR（ypT0yp0）
2. BCS
3. ORR
4. iDFS
5. EFS
6. Security
7. Biomarker detection

Research object： T1c-2N0-1M0 HER2 expression positive in newly treated female patients

ELIGIBILITY:
Inclusion Criteria:

1. Age: Female first-time patients aged 18 and above;
2. Pathological examination confirmed HER2 positive invasive breast cancer; (HER2 positive definition) Further application of in situ hybridization (ISH) for immunohistochemistry (IHC) 3+or IHC 2+HER2 gene amplification, regardless of hormone receptor status (ER and PR);
3. According to the eighth edition of AJCC, the staging is T1c-2N0-1M0, and according to Recipe 1.1, there are At least one measurable lesion;
4. ECOG PS: 0-1 points;
5. The main organ function is normal, which meets the following standards:

1) The standard for blood routine examination must comply with (no blood transfusion or blood products within 14 days, no use of G-CSF) Correction of other hematopoietic stimulating factors:Hb≥100g/L ;ANC≥1.5×109/L；PLT≥100×109/L；2) Biochemical examination must meet the following standards:TBIL≤1×ULN； ALT, AST ≤ 1.5 × ULN; ALP≤2.5×ULN； BUN and Cr ≤ 1.5 × ULN;3) Cardiac ultrasound:Left ventricular ejection fraction (LVEF) ≥ 55%; 6. Women of childbearing age must undergo a pregnancy test (serum) within 7 days before enrollment, and the result is negative Sexual and willing to use appropriate medication during the trial period and within 8 weeks after the last administration of the investigational drug The method of contraception; 7. The subjects voluntarily joined this study, signed an informed consent form, had good compliance, and cooperated with follow-up.

Exclusion Criteria:

1. Have received any form of anti-tumor treatment in the past (chemotherapy, radiotherapy, molecular targeted therapy,...)Endocrine therapy, etc;
2. Simultaneously receiving any other anti-tumor treatment;
3. Bilateral breast cancer, inflammatory breast cancer or occult breast cancer;
4. breast cancer not confirmed by histopathology;
5. Other malignant tumors have appeared within the past 5 years, except for cured cervical cancer in situ;
6. Severe dysfunction of important organs such as heart, liver, and kidney;
7. Unable to swallow, chronic diarrhea, and intestinal obstruction, there are various factors that affect medication administration and absorption factor;
8. Participated in clinical trials of other drugs within 4 weeks prior to enrollment;
9. Individuals with a known history of allergies to the drug components of this protocol; History of immunodeficiency, including HIV Test positive, HCV, active hepatitis B, or other acquired diseases Natural immunodeficiency disease or a history of organ transplantation;
10. Have ever suffered from any heart disease, including: (1) those that require medication or have clinical significance Arrhythmias; (2) Myocardial infarction; (3) Heart failure; (4) Any researcher Other heart diseases deemed unsuitable for participation in this trial;
11. Pregnant and lactating female patients with fertility and positive baseline pregnancy test results Female patients of childbearing age who are unwilling to take effective contraceptive measures throughout the entire trial period Female patients;
12. According to the researcher's judgment, there is a serious threat to patient safety or an impact on patient completion of the study The accompanying diseases studied (including but not limited to severe hypertension that cannot be controlled by medication, severe Diabetes, active infection, etc.);
13. Have a clear history of neurological or psychiatric disorders, including epilepsy or dementia. Researchers believe that Any other circumstances in which the patient is not suitable to participate in this study.

Min Age: 18 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 109 (Estimated)
Dates: Start 2024-07-15 (Estimated); Primary Completion 2026-06-30 (Estimated); Study Completion 2026-12-30 (Estimated)

PRIMARY OUTCOMES:
Follow up on postoperative pathological reports for evaluation for Pathological complete response rate (tpCR: ypT0-is/ypN0) | 18weeks
  Follow up on postoperative pathological reports for evaluation rely onMiller&Payne principles

SECONDARY OUTCOMES:
Objective response rate (ORR) for treatment | At the end of the second cycle (each cycle is 21 or 28 days)]
  The proportion of patients whose tumor volume has shrunk to a predetermined value and can maintain the minimum time limit requirement

IPD SHARING:
Plan to Share IPD: No
Temporarily not sharing, my own ideas